CLINICAL TRIAL: NCT02555995
Title: Assessment of Scan Quality of Sparse OCT Retina Scanner (MimoStudy01)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University Hospital, Zürich (Other); ISS AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-ZH-Nr. 2015-0316
Record Dates: First submitted 2015-09-17; First posted 2015-09-22 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Macular Degeneration
Keywords: AMD; OCT
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All study participants (Experimental): Patient's eyes are OCT-scanned with standard device and investigational device.
  Interventions: Device: OCT scan (as yet unnamed)

INTERVENTIONS:
Device: OCT scan (as yet unnamed) — OCT scan (as yet unnamed) of the eye with investigational device; newly developed sparse OCT retina scanner by Artorg Center Bern and Berner Fachhochschule Biel

SUMMARY:
Optical Coherence Tomography (OCT) is an established non-invasive medical imaging technique ophthalmologists use to diagnose and monitor retinal diseases such as age-related macular degeneration (AMD).

This study assesses the scanning performance of a newly developed sparse OCT retina scanner that is smaller and more compact than most commercially available medical OCT systems. The prototype device was developed at Artorg Center Bern and Berner Fachhochschule Biel.

In this study the device is first tested on human eyes. The scanning performance is compared to a reference device. Additionally patient feedback during the examination is acquired.

The findings of this study are used to improve the software and the ergonomics of the investigational device.

DETAILED DESCRIPTION:
Background

Optical Coherence Tomography (OCT) is an established non-invasive medical imaging technique ophthalmologists use to diagnose and monitor retinal diseases such as age-related macular degeneration (AMD).

This study assesses the scanning performance of a newly developed sparse OCT retina scanner that is smaller and more compact than most commercially available medical OCT systems. The prototype device was developed at Artorg Center Bern and Berner Fachhochschule Biel.

In this study the device is first tested on human eyes. The scanning performance is compared to a reference device. Additionally patient feedback during the examination is acquired.

The findings of this study are used to improve the software and the ergonomics of the investigational device.

Objective

* Comparing scan quality of investigational device to scan quality of reference device.
* Obtaining patient feedback on the examination with investigational device.

Methods

Comparison of OCT scans made with standard device and investigational device.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* German speaking
* Suffering from age-related macular degeneration
* Written informed consent

Exclusion Criteria

* Epilepsy
* Parkinsonian syndrome
* Dementia
* Pregnant women
* Persons using electronic medical aids i.e. hearing aid, pacemaker..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Distance between ILM and RPE (IPD) measurement successful or not. Successful is defined as a) measurement performed/failed, and if performed, b) value obtained within ±10% of value of reference OCT device. | During diagnostic intervention, expected to be ca. 30 minutes on average

SECONDARY OUTCOMES:
Patient comfort during examination | Directly after diagnostic intervention, expected to be ca. 35 minutes on average
  Assessed via interview with patient
Duration of OCT examination with investigational device | Directly after diagnostic intervention, expected to be ca. 35 minutes on average

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Zweifel, MD, Principal Investigator — Augenklinik Universitätspital Zürich; Raphael Sznitman, Study Director — ARTORG, University of Bern
Locations (1):
- Augenklinik Univestitätspital Zürich, Zurich, Canton of Zurich, Switzerland